CLINICAL TRIAL: NCT01162798
Title: Growth of Preterm Infants Consuming Formula
Brief Title: Preterm Infant Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 09.02.US.INF
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Growth; Development; Infant
Keywords: infant formula; premature infants; Growth and Development
MeSH Terms: conditions — Premature Birth | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): commercially available formula
  Interventions: Other: control infant formula
- Test (Experimental): test formula
  Interventions: Other: infant formula

INTERVENTIONS:
Other: infant formula — test infant formula fed to infants until 6 months corrected gestational age
  Other Names: test infant formula
  Arms: Test
Other: control infant formula — commercially available infant formula
  Other Names: commercially available infant formula fed to infants until 6 months corrected gestational age
  Arms: Control

SUMMARY:
The purpose of this study is to assess growth of preterm infants fed a test formula compared to a standard formula up to the first 4 months of corrected gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Born AGA
* Exclusively formula-fed
* 28-34 weeks GA at birth
* Intact GI tract, tolerating full oral feeds
* Expected to be discharged from the hospital within a minimum of 24 hours, maximum of 5 days

Exclusion Criteria:

* Severe respiratory disease defined as needing mechanical ventilation at discharge
* Any significant systemic diseases that could affect growth. This includes cardiac, neurologic, or GI conditions.
* Major congenital malformation, history of GI surgery, severe postnatal complications
* Daily or routine diuretic use at time of discharge
* Receiving more than 10% of daily kcals from food additives such as thickeners
* Currently participating or having participated in another conflicting clinical trial.

Max Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2010-09; Primary Completion 2013-10 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Growth | 4 months
  weight gain assessed monthly

SECONDARY OUTCOMES:
growth, tolerance, morbidity | 6 months
  gains in length and head circumference assessed monthly, tolerance and morbidity throughout study
Total body bone mineral content and density and body composition, protein status, and metabolic markers | corrected term and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard Ziegler, MD, Principal Investigator — University of Iowa
Locations (9):
- United States (9):
  - Children's Hospital & Research Center, Oakland, California
  - Advocate Lutheran Children's Hospital, Park Ridge, Illinois
  - University of Iowa, Iowa City, Iowa
  - Center for Human Nutrition, Omaha, Nebraska
  - Midatlantic Neonatology Associates, Inc, Morristown, New Jersey
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Utah, Dept of Pediatrics, Salt Lake City, Utah
  - VCU Children's Medical Center, Richmond, Virginia